CLINICAL TRIAL: NCT04600440
Title: Convalescent Plasma in the Treatment of Covid-19
Acronym: COP20
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Mona Landin-Olsson, MD Prof, Senior consultant, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Covid convalescent plasma
Record Dates: First submitted 2020-10-20; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Covid-19; Respiratory Insufficiency
Keywords: Covid-19; Convalescent plasma
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma treatment (Experimental): Convalescent plasma 200 ml daily during three days
  Interventions: Biological: Convalescent plasma
- No plasma (No Intervention): Best conventional treatment

INTERVENTIONS:
Biological: Convalescent plasma — Plasma donated from patients recovered from Covid-19 and having high titres of antibodies
  Arms: Plasma treatment

SUMMARY:
One hundred patients hospitalized and in need of oxygen treatment due to Covid-19 should be randomized and 50% treated with 200 ml convalescent plasma x 3 and 50% given ordinary treatment.

Primary outcome is number of days the patients need oxygen within 28 days from inclusion.

Secondary outcome is number of days in hospital, number of days in respirator and mortality.

Side effects of treatment is monitored.

DETAILED DESCRIPTION:
Subjects with previous verified COVID-19 are asked to donate plasma 14 days or later after recovery. IgG antibodies against Covid-19 are measured and only subjects with high titers are accepted. Plasmaphereses is done and up to 600 ml plasma is drawn and aliquoted in 200 ml portions.

Patients with acute respiratory symptoms, verified Covid-19, hospitalized and in need of oxygen treatment are asked to participate in the study. The patients are randomized 50/50 to get either convalescent plasma or routine treatment without plasma. The patients randomized to get plasma will have infusion of 200 ml blood group compatible convalescent plasma daily during three days from different donors.

The clinical course will be carefully monitored and days with oxygen requirement will be compared between the groups. Secondary clinical outcomes as mortality, need of assisted ventilation, total days in hospital and side effects to treatment will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of Covid-19
* <94% oxygen saturation
* willingness to participate
* ability to sign informed consent

Exclusion Criteria:

* unability to understand information and sign informed consent
* immunosuppressed patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of days in need of oxygen | 28 days
  Number of days in need of oxygen within 28 days from inclusion

SECONDARY OUTCOMES:
Number of days before discharge from hospital | 3 months
  number of days before discharge from hospital
Mortality within 3 months | 3 months
  death of patient
Number of days before need of assisted ventilation | 28 days
  number of days before need of assisted ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Mona Landin-Olsson, MD, Prof, Principal Investigator — Skane University Hospital; Maria N Lundgren, MD, Study Chair — Skane University Hospital
Locations (1):
- Skåne University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Holm K, Lundgren MN, Kjeldsen-Kragh J, Ljungquist O, Bottiger B, Wiken C, Oberg J, Fernstrom N, Rosendal E, Overby AK, Wigren Bystrom J, Forsell M, Landin-Olsson M, Rasmussen M. Convalescence plasma treatment of COVID-19: results from a prematurely terminated randomized controlled open-label study in Southern Sweden. BMC Res Notes. 2021 Dec 4;14(1):440. doi: 10.1186/s13104-021-05847-7. PMID 34863304